CLINICAL TRIAL: NCT06741904
Title: Noninvasive Methods for Predicting the Occurrence of Decompensation in Chronic Liver Disease: a Prospective, Observational, Multicenter Study
Brief Title: Non-invasive Methods for Predicting Decompensation of Chronic Liver Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-427
Record Dates: First submitted 2024-12-04; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Chronic Liver Disease and Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preliminary studies have suggested that non-invasive methods can not only be applied to CSPH but also to predict the risk of decompensation in cirrhosis. However, there is a lack of clinical evidence, and more research is needed to provide such evidence. Especially in China, where the etiology of cirrhosis is prevalent, there is a large population of patients with hepatitis B cirrhosis undergoing antiviral treatment. Exploring the value of non-invasive methods in predicting decompensation events in these patients can not only expand the clinical application of non-invasive methods but also provide effective non-invasive screening and management strategies for patients with cirrhosis at different risk levels.

Primary Objective: The main purpose of this study is to evaluate the predictive effectiveness of non-invasive methods (based on liver and spleen stiffness) for the occurrence of decompensation in chronic liver disease (CLD).

Secondary Objectives: To establish different predictive models for the occurrence of decompensation in CLD and to assess their predictive effectiveness as non-invasive methods for decompensation in CLD.

Approximately 2334 individuals will participate in this study at 17 different health care Setting.The study will last for 4 years, including 1 year of enrollment and 3 years of follow-up. Patients will be seen at 6-month intervals, and all examination results of patients as well as decompensation events, liver cancer, and death will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years and under 80 years; ② Underlying chronic liver disease (etiology not specified);

  * Liver stiffness measurement (LSM) greater than 10 kPa or cirrhosis (diagnosed by imaging or histology);

    * Voluntarily signing an informed consent form.

Exclusion Criteria:

* Have undergone orthotopic liver transplantation or Transjugular Intrahepatic Portosystemic Shunt (TIPS) procedure;

  * History of liver cancer or other types of cancer diagnosed in the past or currently;

    * Acute or chronic portal vein thrombosis; ④ History of splenectomy or splenic embolization; ⑤ Currently in a decompensated stage (with complications such as variceal bleeding, moderate to severe ascites, hepatic encephalopathy, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Liver Disease
Sampling Method: Non-Probability Sample
Enrollment: 2334 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Decompensation events | Patients were followed from the time of enrollment for a maximum of 3 years
  Decompensated events included ascites, variceal bleeding, and hepatic encephalopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dajti E, Ravaioli F, Zykus R, Rautou PE, Elkrief L, Grgurevic I, Stefanescu H, Hirooka M, Fraquelli M, Rosselli M, Chang PEJ, Piscaglia F, Reiberger T, Llop E, Mueller S, Marasco G, Berzigotti A, Colli A, Festi D, Colecchia A; Spleen Stiffness-IPD-MA Study Group. Accuracy of spleen stiffness measurement for the diagnosis of clinically significant portal hypertension in patients with compensated advanced chronic liver disease: a systematic review and individual patient data meta-analysis. Lancet Gastroenterol Hepatol. 2023 Sep;8(9):816-828. doi: 10.1016/S2468-1253(23)00150-4. Epub 2023 Jul 18. PMID 37478880